CLINICAL TRIAL: NCT01184521
Title: Use of the Masimo Rainbow SET Pulse CO-Oximeter in Patients Undergoing Isovolemic Hemodilution
Brief Title: Masimo CO-Oximeter Study
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB10-00364
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulse CO-oximeter

SUMMARY:
This is a study to evaluate the accuracy of the Masimo Rainbow SET Pulse CO-Oximeter in monitoring the hemoglobin levels of patients undergoing isovolemic hemodilution.

ELIGIBILITY:
Inclusion Criteria:

* Any subject that is scheduled to have isovolemic hemodilution

Exclusion Criteria:

* Anything that prevents a subject from having isovolemic hemodilution

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring isovolemic hemodilution during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
hemoglobin value | 1 Day (day of surgery)
  The accuracy of the hemoglobin value from the Masimo pulse oximeter during isovolemic hemodilution.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States